CLINICAL TRIAL: NCT02295735
Title: A Randomized Controlled Parallel-group Trial to Investigate the Effectiveness of Two Silicone Dressings for Sacral and Heel Pressure Ulcer Prevention Compared to no Dressings
Brief Title: Effectiveness of Two Silicone Dressings for Sacral and Heel Pressure Ulcer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PD Dr. Jan Kottner (Other)
Responsible Party: Sponsor-Investigator, PD Dr. Jan Kottner, PD Dr. rer cur, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRC-PU-A-16
Record Dates: First submitted 2014-11-10; First posted 2014-11-20 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Pressure Ulcer
Keywords: Skin, safety, wounds, intensive care
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepilex® Border (Experimental): If a patient is assigned to the intervention group the dressings Mepilex® Border Sacrum and Mepilex® Border Heel will be applied onto the respective intact skin areas in addition to standard pressure ulcer prevention
  Interventions: Device: Mepilex® Border Sacrum and Mepilex® Border Heel
- Control (No Intervention): Standard pressure ulcer prevention according to hospital standard

INTERVENTIONS:
Device: Mepilex® Border Sacrum and Mepilex® Border Heel
  Arms: Mepilex® Border

SUMMARY:
The aim of this randomized controlled trial is to test the efficacy of preventive dressings for pressure ulcer prevention.

DETAILED DESCRIPTION:
Patients of intensive acute care and residents of institutional long-term care facilities are at high risk for developing pressure ulcers (PUs). PU standard prevention includes repositioning, early mobilization and the use of special support surfaces. The use of prophylactic dressings might reduce friction and shear forces and/or modify the microclimate of the skin and might therefore protect the skin and underlying tissues from pressure/deformation injury. The primary objective of this study is to determine if preventive silicone dressings (Mepilex® border) applied to the heels and to the sacrum in addition to PU standard prevention reduces PU incidence category II, III, IV, and deep tissue injury compared to PU standard alone in at risk hospital patients.

ELIGIBILITY:
* Major trauma patients and/or critically ill patients (e.g. with cardiac arrest) admitted to the emergency department and being transferred and/or admitted directly to a surgical or internal ICU
* Being at "high" or "very high" PU risk according to the Charité PU prevention standard:

  - Category 3 (= partly care dependent/limited mobility in bed), 4A (= care depended, limited mobility in bed), 4B (= totally immobile) according to the Jones classification modified by Charité
* Expected minimum length of stay at least three days
* Informed consent (or by legal representative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kottner, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a tertiary care hospital from June 2015 to July 2018 at the Charite Universitaetsmedizin Berlin, Germany. Patients were recruited from seven ICUs.
  In total, 7575 ICU patients were screened for eligibility and 475 ICU patients were included.
Groups:
- Intervention Group: For patients in the intervention group, dressings were applied on both heels (Mepilex Border Heel, Moelnlycke Health Care, Gothenburg, Sweden) and on the sacral areas (Mepilex Border Sacrum, Moelnlycke Health Care) according to manufacturers instructions in addition to the standard care.
- Control Group: Standard pressure ulcer prevention according to hospital standard
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 238 | 237
Completed | 212 | 210
Not Completed | 26 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 212 | 210 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (15.6) | 63.1 (15.2) | 63.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 82 | 146
  Male | 148 | 128 | 276
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 212 | 210 | 422
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — Population: The analyzed Population differs from the Overall due to missing data
  kg/m²
    number analyzed (Participants) | 199 | 202 | 401
    (all) | 26.4 (4.9) | 26.6 (4.8) | 26.5 (4.9)
Braden scale score [Mean (Standard Deviation); unit: units on a scale] — The Braden scale is a standardized six item Pressure ulcer risk assessment instrument with scores ranging from 6 (= high Pressure ulcer risk) to 23 (= no Pressure ulcer risk).
  units on a scale | 8.9 (1.4) | 9.0 (1.6) | 8.9 (1.5)
High Pressure ulcer risk [Count of Participants; unit: Participants] — According to Hospital Standard
  Participants | 20 | 19 | 39
Very high Pressure ulcer risk [Count of Participants; unit: Participants] — According to Hospital Standard
  Participants | 192 | 191 | 383

OUTCOME MEASURES:

1. Primary Outcome: Number of Pressure Ulcers Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum (Proportion)
Description: The primary outcome was the cumulative incidence of Pressure ulcer category II, III, IV, unstageable and DTI at heels or sacrum. Pressure ulcers were categorized according to the NPUAP/EPUAP 2014 classification System. The occurrence of a new pressure ulcer of any category was assessed and documented daily during the study period. The Categories are defined as follows: Category I (nonblanchable erythema); Category II (Partial thickness Skin loss); Category III (Full Thickness Skin loss); Category IV (Full Thickness tissue loss); Unstageable (Depth unknown); Deep tissue injury (suspected Deep tissue injury, Depth unknown)
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: Pressure ulcer
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
Pressure ulcer | 6 | 22

2. Secondary Outcome: Density Rate of Pressure Ulcers Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum (Proportion Per 1000 Bed Days, Rate)
Description: The Incidence density of Pressure Ulcer category II, III, IV, unstageable and DTI at heels or sacrum was measured. Pressure ulcer were categorized according to the NPUAP/EPUAP 2014 classification system. The occurrence of a new Pressure ulcer of any category was assessed and documented daily during the study period. The Categories are defined as follows: Category I (nonblanchable erythema); Category II (Partial thickness Skin loss); Category III (Full Thickness Skin loss); Category IV (Full Thickness tissue loss); Unstageable (Depth unknown); Deep tissue injury (suspected Deep tissue injury, Depth unknown)
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: Proportion developed / 1000 bed days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
Proportion developed / 1000 bed days | 7.8 | 30.5

3. Secondary Outcome: Number of Pressure Ulcer Category I (Non-blanchable Erythema) II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum (Proportion)
Description: The the cumulative incidence of Pressure ulcer category I, II, III, IV, unstageable and DTI at heels or sacrum. Pressure ulcer were categorized according to the NPUAP/EPUAP 2014 classification system. The occurrence of a new Pressure ulcer of any category was assessed and documented daily during the study period. The Categories are defined as follows: Category I (nonblanchable erythema); Category II (Partial thickness Skin loss); Category III (Full Thickness Skin loss); Category IV (Full Thickness tissue loss); Unstageable (Depth unknown); Deep tissue injury (suspected Deep tissue injury, Depth unknown)
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: Pressure ulcer
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
Pressure ulcer | 6 | 28

4. Secondary Outcome: Number of Pressure Ulcers Category I (Non-blanchable Erythema) II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum (Proportion Per 1000 Bed Days, Rate)
Description: The Incidence density of Pressure Ulcer category I, II, III, IV, unstageable and DTI at heels or sacrum was measured. Pressure ulcer were categorized according to the NPUAP/EPUAP 2014 classification system. The occurrence of a new Pressure ulcer of any category was assessed and documented daily during the study period. The Categories are defined as follows: Category I (nonblanchable erythema); Category II (Partial thickness Skin loss); Category III (Full Thickness Skin loss); Category IV (Full Thickness tissue loss); Unstageable (Depth unknown); Deep tissue injury (suspected Deep tissue injury, Depth unknown)
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: Proportion developed / 1000 bed days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
Proportion developed / 1000 bed days | 8.0 | 37.6

5. Secondary Outcome: Number of Preventive Sacrum Dressings Used for Pressure Ulcer Prevention
Description: Number of preventive sacrum dressings used for pressure ulcer prevention
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: Dressings
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
Dressings | 1050 | 0

6. Secondary Outcome: Numbers of Support Surface Used for Pressure Ulcer Prevention (Total)
Description: Support surface categories were recorded. Please see the different types in the Outcome measure data table
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: number of support surfaces used
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
number of support surfaces used
  Total numbers of support surfaces used | 212 | 209
  non-powered systems | 149 | 117
  powered - alternating Systems | 79 | 85
  powered - low-air-loss Systems | 1 | 5
  other | 3 | 2

7. Secondary Outcome: Time to Pressure Ulcer Development of Pressure Ulcers Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum
Description: • Time to Pressure ulcer development in days
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
days | 10.8 (10.1) | 13.5 (13.8)

8. Secondary Outcome: Number of Preventive Heel Dressings Used for Pressure Ulcer Prevention
Description: Number of preventive heel dressings used for pressure ulcer prevention
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Number; unit: Dressings
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
Dressings | 2260 | 0

9. Secondary Outcome: Time to Pressure Ulcer Development of Pressure Ulcers Category I, II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum
Description: • Time to Pressure ulcer development in days
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
days | 10.8 (10.1) | 13.2 (12.4)

10. Secondary Outcome: Event Free Survival Time of Pressure Ulcers Category II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum (Days, Kaplan Meier Analysis)
Description: • Estimation of the Survival function and measure of the length of time the ICU patients remained Pressure ulcer free in days
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Mean (Standard Error); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
days | 60.7 (4.1) | 89.0 (9.8)

11. Secondary Outcome: Event Free Survival Time of Pressure Ulcers Category I, II, III, IV, Unstageable, Deep Tissue Injury (DTI) at Heels and/or Sacrum (Days, Kaplan Meier Analysis)
Description: as for outcome 10
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Mean (Standard Error); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
days | 60.7 (4.1) | 54.6 (9.1)

12. Secondary Outcome: Follow up Period of Included ICU Patients (Days)
Description: Follow up period of included ICU patients in mean (days)
Time Frame: Duration of hospital stay, an average of 12.6 (SD +/-12.7) days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 210
days | 11.0 (10.3) | 14.3 (14.6)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded every day until the Patient was discharged from the Hospital,an average of 12.6 (SD +/-12.7) days
Description: Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device.
  Note: This definition includes events related to the investigational medical device or the comparator. This definition includes events related to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/210
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/210
Other Adverse Events (participants affected / at risk) | 2/212 | 0/210
OTHER ADVERSE EVENTS (reported when occurring in more than 0.47% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=212) | Control Group (N=210)
Burning pain and warm sensation under the sacral dressing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peeling of the outer layers of the skin under the sacral dressing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02295735/Prot_SAP_000.pdf